CLINICAL TRIAL: NCT03722537
Title: Osteochondral Allograft in the Surgical Treatment of Basal Joint Arthritis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative changes
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAS2615
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Basal Joint Arthritis
Keywords: Allograft; Osteochondral Allograft; Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligament Reconstruction Tendon Interposition (LRTI) (Active Comparator): Selected randomly, 100 patients will receive this treatment. During the LRTI (standard of care procedure), the arthritic bone that the thumb rests on (the trapezium) is removed. A small cut is made in the forearm to release a tendon, which is moved to the base of the thumb to fill in the area from which the trapezium bone was removed. A small suture anchor is then placed into a thumb bone which holds everything together.
  Interventions: Procedure: Ligament Reconstruction Tendon Interposition
- Osteochondral Allograft (Experimental): Selected randomly,100 patients will receive this treatment. In this procedure, the arthritic bone that the thumb rests on (the trapezium) is removed and replaced with femoral trochlear osteochondral allograft that is designed to be similar in morphology to the human trapezium articular surface, known as the 'Cartibend©' .
  Interventions: Procedure: Osteochondral Allograft

INTERVENTIONS:
Procedure: Osteochondral Allograft — The arthritic bone that the thumb rests on (the trapezium) is removed and replaced with femoral trochlear osteochondral allograft that is designed to be similar in morphology to the human trapezium articular surface.
  Other Names: Cartibend
  Arms: Osteochondral Allograft
Procedure: Ligament Reconstruction Tendon Interposition — During the LRTI, the arthritic bone that the thumb rests on (the trapezium) is removed. A small cut is made in the forearm to release a tendon, which is moved to the base of the thumb to fill in the area from which the trapezium bone was removed. A small suture anchor is then placed into a thumb bone which holds everything together.
  Arms: Ligament Reconstruction Tendon Interposition (LRTI)

SUMMARY:
This is a study comparing the current standard of care surgical treatment to a newer surgical procedure involving the implantation of osteochondral allograft at the base of the thumb. Patients will be followed at 1, 3, 6 months and 1 year post-operatively.

DETAILED DESCRIPTION:
Basal joint arthritis of the thumb is a common condition associated with considerable morbidity. Many non-operative and operative treatments have been described, but few multicenter prospective evidence based trials exist comparing standard treatments. This continuing search for consensus and improvement of best clinical practice has been reviewed in a thorough meta-analysis of operative treatments for basal joint arthritis. Operative treatments range from osteotomy, partial or complete trapeziectomy with or without reconstruction of the ligaments, tendon interposition to arthrodesis, however the functional outcome varies. Allograft has been previously described in joint replacement / prosthetic implantation surgery in other areas of the body, however not in the thumb. The purpose of this study is to investigate using osteochondral allograft in the surgical intervention phase of treatment for patients with basal joint arthritis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Indicated for operative management of basal joint arthritis

Exclusion Criteria:

* Pregnant women/fetuses/neonates, prisoners
* Previously operated on for treatment of basal joint arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Score on the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire | Up to 1 year post-operatively
  The DASH (Disabilities of the Arm, Shoulder, and Hand) is a 30-item questionnaire that includes 21 physical function items, 6 symptom items, and 3 social/role function items used to evaluate a patient's ability to perform upper extremity activities. Higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability. The score on both test ranges from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
Score on the Thumb Disability Exam (TDX) | Up to 1 year post-operatively
  The TDX is a questionnaire that measures changes in thumb function and pain, specifically for those with basal joint arthritis.The TDX is scored on a scale of 0 to 100, with a higher score indicating a greater degree of disability in the thumb.
Visual Analog Scale for pain (VAS) | Up to 1 year post-operatively
  The VAS is a validated technique that measures acute and chronic pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Melvin P Rosenwasser, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No